CLINICAL TRIAL: NCT06609460
Title: A Phase 2b Randomized, Double-blind, Placebo-controlled, Multicenter Dose Ranging Study to Evaluate Efficacy and Safety of CD388, a Novel Long-acting Antiviral Conjugate, for the Prevention of Influenza in Subjects Not at Risk for Influenza Complications
Brief Title: Study of CD388 for the Prevention of Influenza in Subjects Not at Risk for Influenza Complications
Acronym: NAVIGATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CD388.SQ.2.05
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CD388 Low Dose (Experimental): Participants are randomized to receive a low dose of CD388 by SQ injection. Participants are randomized at a 1:1:1:1 ratio across the 4 arms.
  Interventions: Combination Product: CD388 Injection
- CD388 Medium Dose (Experimental): Participants are randomized to receive a medium dose of CD388 by SQ injection. Participants are randomized at a 1:1:1:1 ratio across the 4 arms.
  Interventions: Combination Product: CD388 Injection
- CD388 High Dose (Experimental): Participants are randomized to receive a high dose of CD388 by SQ injection. Participants are randomized at a 1:1:1:1 ratio across the 4 arms.
  Interventions: Combination Product: CD388 Injection
- Placebo (Placebo Comparator): Participants are randomized to receive placebo by SQ injection. Participants are randomized at a 1:1:1:1 ratio across the 4 arms.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: CD388 Injection — CD388 liquid for injection
  Arms: CD388 High Dose; CD388 Low Dose; CD388 Medium Dose
Combination Product: Placebo — Placebo to match
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of CD388 in preventing symptomatic laboratory-confirmed influenza infections, as compared to placebo, and to select a dose of CD388 that is effective in preventing the same, when administered as a single dose via 3 subcutaneous (SQ) injections to adult participants in stable health, and to evaluate the safety and tolerability of CD388, as compared to placebo.

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, double-blind, placebo-controlled, parallel-group, multicenter dose selection study to evaluate the efficacy, safety, and tolerability of 3 dose levels of CD388 administered as a single dose via 3 SQ injections in adult participants who are not at risk of developing complications from influenza.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent and comply with scheduled visits, laboratory tests, and other study procedures.
2. Males and females 18 to less than 64 years of age.
3. In the Investigator's clinical judgment, is in stable health at the time of screening and randomization. Participants may not have underlying hematologic, oncologic, renal, autoimmune, and/or cardiopulmonary illnesses or be considered at risk of developing complications from influenza infection per the CDC guidelines (chronic obstructive pulmonary disease [COPD], asthma, immune compromised current cancer [except non-melanomatous skin cancer], or diabetes). Subjects will be included on the basis of medical history and vital signs taken between signing of the informed consent and randomization.
4. Body mass index (BMI; calculated as weight in kilograms [kg] divided by height in meters [m] squared) of 18.0 kg/m^2 to 35.0 kg/m^2 (inclusive).
5. Women of childbearing potential (WOCBP) must:

   1. Have a negative pregnancy test (beta-human chorionic gonadotropin [β-hCG]) at screening, AND
   2. Be practicing a highly effective, preferably user-independent method of contraception (failure rate of less than 1 percent per year when used consistently and correctly) from ≥2 weeks prior to randomization and agrees to remain on a highly effective method from Day 1 until 32 weeks after study drug administration, the end of relevant systemic exposure. The Investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the day of administration of study drug.

   A woman is considered of childbearing potential (i.e., fertile) following menarche and until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
6. Female participants must agree not to donate or freeze eggs (ova, oocytes) for future use for the purposes of assisted reproduction from Day 1 until 32 weeks after study drug administration.
7. Male participants must wear a condom when engaging in any activity that allows for passage of ejaculate to another person from Day 1 until 32 weeks after study drug administration. Male participants should also be advised of the benefit for a female partner to additionally use a highly effective method of contraception, as condoms could break or leak.

   Note: Contraceptive (birth control) use by participants should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies.
8. Male participants must agree not to donate sperm from Day 1 until 32 weeks after study drug administration.
9. Participant agrees not to donate blood from Day 1 until 32 weeks after study drug administration.
10. Must be able to read, understand, and complete questionnaires in the electronic diary (eDiary), work with smartphones/tablets/computers, and be willing and able to adhere to the prohibitions and restrictions specified in this protocol. If an appropriate language version is not available for the eDiary assessments, the participant should not be enrolled.
11. Must be willing to provide verifiable identification, has means to be contacted, and is able to contact the Investigator/study site and communicate reliably during participation in the study.

Exclusion Criteria:

1. Known or suspected allergy or history of anaphylaxis or other serious adverse reactions to zanamivir (following administration of inhaled or intravenous formulations), monoclonal antibodies (including crystallizable fragment [Fc] domains), or any of the components of CD388 or placebo.
2. Have been diagnosed with influenza (i.e., with medical history [including verbal] of influenza) within the past 6 months prior to randomization.
3. Has received the current seasonal influenza vaccine prior to screening or is planning to receive the seasonal vaccine during trial participation.
4. Has an acute illness (including acute respiratory illnesses) or body temperature ≥38.0ºC (≥100.4 degrees Fahrenheit [ºF]) within 7 days prior to study drug administration (Note: Enrollment at a later date, subsequent to resolution [within the screening period] is permitted).
5. Has had close contact (including household contacts) with someone with laboratory-confirmed influenza or with someone who has been treated with antiviral therapies for influenza within the past 7 days prior to randomization.
6. Has had close contact (including household contacts) with someone with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection or coronavirus disease 2019 (COVID-19) as defined by the US CDC or has had a positive SARS-CoV-2 test within 10 days prior to screening. Please note SARS-CoV-2 testing is NOT required during screening.
7. Has a serious and/or clinically unstable condition such as psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior, Alzheimer's disease, or any other condition for which, in the opinion of the Investigator, participation would not be in the participant's best interest or that could prevent, confound, or limit the protocol-specified assessments.
8. Any history of alcohol or drug abuse within the past 2 years or a positive urine drug screen for drugs of abuse (other than tetrahydrocannabinol [THC]) at screening or Day 1. Note: urine drug screen that is positive for a medication prescribed for treatment of ongoing condition is not exclusionary.
9. Had major surgery (e.g., major cardiopulmonary or abdominal operations) per Investigator judgment within 4 weeks prior to randomization, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to participate in the study.
10. Screening ECG findings of prolonged QT interval corrected for heart rate using Fridericias formula (QTcF) (greater than 450 milliseconds [msec] in males or greater than 470 msec in females), prolonged PR interval (greater than 220 msec), second- or third-degree heart block, or other clinically significant dysrhythmias.
11. At the time of screening, any finding that may significantly increase the risk of participation in the study, affect the ability to participate in the study, or impair interpretation of the study data.
12. Current or planned participation in another clinical study where study intervention is being administered while participating in the current study. Note: Concurrent enrollment is allowed during the follow-up phase of the other clinical study or in case the study intervention in the other clinical study is a marketed product already approved for another indication - exception being if the other study requires study interventions that could affect the safety assessments of the present study (e.g., clinical laboratory tests).
13. [Exclusion criterion #13 removed during Amendment 1.1-US; placeholder remains to retain numbering of the remaining original exclusion criteria.]
14. Prior receipt within the past 30 days or 5 half-lives (whichever is longer) or anticipated receipt of any drug, vaccine, or other biologic agent (e.g., monoclonal antibodies) administered for the prevention or treatment of influenza.
15. Prior receipt of any experimental drug, vaccine, or biologic agent within the past 90 days or 5 half-lives (whichever is longer).
16. Contraindication to SQ injections and blood draws (e.g., bleeding disorders).
17. Has donated ≥450 mL of blood product (1 unit) for any reason within 30 days of screening or plans to donate blood product during the study.
18. Currently pregnant or breastfeeding, intends to become pregnant or breastfeed, or has a positive pregnancy test during the screening period.
19. Has direct involvement in the proposed study or other studies under the direction of the Investigator, sub-investigators, or study site; is a family member of an individual with such direct involvement; or is an employee of the Sponsor.
20. In the opinion of the Investigator, is unlikely to adhere to the requirements of the study.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5071 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Protocol-defined Influenza-like Illness (ILI) Occurring ≥7 Days after and up to 24 Weeks after Administration of Study Drug | From Day 8 up to 24 weeks after study drug dosing
  Percentage of participants experiencing protocol-defined ILI occurring after administration of CD388, with central laboratory-confirmed reverse-transcriptase polymerase chain reaction positive (RT-PCR+) influenza infection based on the nasopharyngeal (NP) swab result, as compared to placebo.
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) after Administration of Study Drug | From Day 1 through Day 197/End of Study (EOS) after study drug dosing
  Safety and tolerability of CD388, as compared to placebo, will be evaluated by assessing the number of participants with incidences of TEAEs following the administration of study drug. TEAEs include but are not limited to adverse events (AEs), serious adverse events (SAEs), injection site reactions (ISRs), and any potentially clinically significant changes from baseline seen in vital signs, 12-lead electrocardiograms (ECGs), and clinical laboratory parameters.

SECONDARY OUTCOMES:
Percentage of Participants Experiencing Protocol-defined ILI Occurring ≥7 Days after and up to 28 Weeks after Administration of Study Drug | From Day 8 up to 28 weeks after study drug dosing
  Percentage of participants experiencing protocol-defined ILI occurring after administration of CD388, with central laboratory-confirmed RT-PCR+ influenza infection based on the NP swab result, as compared to placebo.
Percentage of Participants Experiencing Protocol-defined ILI (as in Primary Endpoint 1) Except with a Lower Threshold for New Onset of Fever | From Day 8 up to 24 weeks after study drug dosing
  Percentage of participants experiencing protocol-defined ILI occurring after administration of CD388, with central laboratory-confirmed RT-PCR+ influenza infection based on the NP swab result, as compared to placebo. New onset of fever is defined as oral temperature ≥37.2 degrees Celsius (°C). Respiratory symptoms are influenza-associated and as described in the protocol. Onset events include those occurring ≥7 days after and up to 24 weeks following study drug administration.
Percentage of Participants Experiencing Protocol-defined ILI (as in Primary Endpoint 1) Except the Influenza Infection is Based on the Midturbinate (MT) Swab Result | From Day 8 up to 24 weeks after study drug dosing
  Percentage of participants experiencing protocol-defined ILI occurring after administration of CD388, with the influenza infection based on the MT swab result, as compared to placebo.
Percentage of Participants Experiencing an Influenza Infection AND New Onset of Fever AND New Onset of ≥2 Respiratory Symptoms after Administration of Study Drug | From Day 8 up to 24 weeks after study drug dosing
  Percentage of participants experiencing a central laboratory-confirmed RT-PCR+ influenza infection based on the NP swab result (first occurrence only) occurring after administration of CD388, as compared to placebo. New onset of fever is defined as oral temperature ≥37.8°C. Respiratory symptoms are influenza-associated and as described in the protocol. Onset events include those occurring ≥7 days after and up to 24 weeks following study drug administration.
Percentage of Participants Experiencing an Influenza Infection AND New Onset of ≥2 Respiratory Symptoms after Administration of Study Drug | From Day 8 up to 24 weeks after study drug dosing
  Percentage of participants experiencing a central laboratory-confirmed RT-PCR+ influenza infection based on the NP swab result (first occurrence only) occurring after administration of CD388, as compared to placebo. Respiratory symptoms are influenza-associated and as described in the protocol. Onset events include those occurring ≥7 days after and up to 24 weeks following study drug administration.
Percentage of Participants Experiencing an Influenza Infection AND New Onset of ≥1 Respiratory Symptom AND New Onset of ≥1 Systemic Symptom after Administration of Study Drug | From Day 8 up to 24 weeks after study drug dosing
  Percentage of participants experiencing a central laboratory-confirmed RT-PCR+ influenza infection based on the NP swab result (first occurrence only) occurring after administration of CD388, as compared to placebo. Respiratory symptoms are influenza-associated and as described in the protocol. Onset events include those occurring ≥7 days after and up to 24 weeks following study drug administration.
Percentage of Participants Experiencing an Influenza Infection, AND New Onset of ≥2 Respiratory Symptoms, OR ≥1 Respiratory Symptom AND New Onset of ≥1 Systemic Symptom, after Administration of Study Drug | From Day 8 up to 24 weeks after study drug dosing
  Percentage of participants experiencing a central laboratory-confirmed RT-PCR+ influenza infection based on the NP swab result (first occurrence only) occurring after administration of CD388, as compared to placebo. Respiratory symptoms are influenza-associated and as described in the protocol. Onset events include those occurring ≥7 days after and up to 24 weeks following study drug administration.
Percentage of Participants Experiencing an Influenza Infection AND New Onset of Fever, AND New Onset of ≥2 Respiratory Symptoms, OR New Onset of ≥1 Respiratory Symptom Plus New Onset of ≥1 Systemic Symptom, after Administration of Study Drug | From Day 8 up to 24 weeks after study drug dosing
  Percentage of participants experiencing a central laboratory-confirmed RT-PCR+ influenza infection (first occurrence only) from either the self-collected MT swab (collected prior to the initiation of any antiviral treatment) or the NP swab collected by a health professional, occurring after administration of CD388, as compared to placebo. New onset of fever is defined as oral temperature ≥38°C. Respiratory symptoms are influenza-associated and as described in the protocol. Onset events include those occurring ≥7 days after and up to 24 weeks following study drug administration.
Severity (as Composite Symptom Score) of Participant Reported Influenza-like Symptoms as Based on the Self-reported Responses to the Respiratory Infection Intensity and Impact Questionnaire (RiiQ™) Symptom Scale | On Day 1 (pre-dose baseline); and then once daily from the time the participant triggers an ARI Alert in the eDiary until the ARI episode is resolved for a maximum of 29 days per ARI episode, up to 28 weeks after study drug dosing
  Evaluation of the severity (defined as the composite symptom score) of participant reported influenza-like symptoms as based on the self-reported responses to the RiiQ™ Symptom Scale (scored as 0 = none, 1 = mild, 2 = moderate, and 3 = severe) as presented in the participant eDiary. The composite symptom score is defined as the mean of the scores of the non-missing influenza symptoms for each time point. From the time the participant triggers an Acute Respiratory Infection (ARI) Alert in the eDiary until the ARI episode is resolved (defined as 2 consecutive days where all influenza-associated symptoms on the RiiQ™ Symptom Scale have returned to the same severity level as reported at baseline or lower), the participant will complete the RiiQ™ Symptom Scale in the eDiary for a maximum of 29 days, per ARI episode.
Severity (as Area Under the Curve [AUC]) of Participant Reported Influenza-like Symptoms as Based on the Self-reported Responses to the RiiQ™ Symptom Scale | On Day 1 (pre-dose baseline); and then once daily from the time the participant triggers an ARI Alert in the eDiary until the ARI episode is resolved for a maximum of 29 days per ARI episode, up to 28 weeks after study drug dosing
  Evaluation of the severity (presented as AUC) of participant reported influenza-like symptoms as based on the self-reported responses to the RiiQ™ Symptom Scale (scored as 0 = none, 1 = mild, 2 = moderate, and 3 = severe) as presented in the participant eDiary. AUC will be based on scores of the non-missing influenza symptoms for each time point. From the time the participant triggers an Acute Respiratory Infection (ARI) Alert in the eDiary until the ARI episode is resolved (defined as 2 consecutive days where all influenza-associated symptoms on the RiiQ™ Symptom Scale have returned to the same severity level as reported at baseline or lower), the participant will complete the RiiQ™ Symptom Scale in the eDiary for a maximum of 29 days, per ARI episode.
Duration (as Time to Symptom Resolution) of Participant Reported Influenza-like Symptoms as Based on the Self-reported Responses to the RiiQ™ Symptom Scale | On Day 1 (pre-dose baseline); and then once daily from the time the participant triggers an ARI Alert in the eDiary until the ARI episode is resolved for a maximum of 29 days per ARI episode, up to 28 weeks after study drug dosing
  Evaluation of the duration (defined as the time from the first report of influenza-associated symptoms to resolution) of participant reported influenza-like symptoms as based on the self-reported responses to the RiiQ™ Symptom Scale (scored as 0 = none, 1 = mild, 2 = moderate, and 3 = severe) as presented in the participant eDiary. From the time the participant triggers an Acute Respiratory Infection (ARI) Alert in the eDiary until the ARI episode is resolved (defined as 2 consecutive days where all influenza-associated symptoms on the RiiQ™ Symptom Scale have returned to the same severity level as reported at baseline or lower), the participant will complete the RiiQ™ Symptom Scale in the eDiary for a maximum of 29 days, per ARI episode.
Trough Plasma Concentration at 24 Weeks (C[trough24w]) Following Administration of CD388 | Based on sampling done at onsite visits on Day 85 (±3 days) and Day 197/EOS (±7 days)
  Evaluation of the trough plasma concentration at 24 weeks (C[trough24w]) after study drug dosing. PK parameters will be assessed in approximately 120 participants at designated sites only.
Maximum Plasma Concentration (C[max]) Following Administration of CD388 | At onsite visits done on Day 8, Day 29, and Day 85 (each ±3 days) and on Day 197/EOS (±7 days)
  Evaluation of the maximum plasma concentration (C[max]) after study drug dosing. PK parameters will be assessed in approximately 120 participants at designated sites only.
Area Under the Plasma Concentration-Time Curve (AUC) Following Administration of CD388 | At onsite visits done on Day 8, Day 29, and Day 85 (each ±3 days) and on Day 197/EOS (±7 days)
  Evaluation of the area under the plasma concentration-time curve (AUC) after study drug dosing. PK parameters will be assessed in approximately 120 participants at designated sites only.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Davarpanah, MD, JD, Study Director — Cidara Therapeutics Inc.
Locations (57):
- United States (56):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Fiel Family and Sports Medicine/CCT Research, Tempe, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Velocity Clinical Research - Huntington Park, Huntington Park, California
  - Velocity Clinical Research - San Diego, La Mesa, California
  - Catalina Research Institute, LLC, Montclair, California
  - Profound Research LLC, Oceanside, California
  - Acclaim Clinical Research, San Diego, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Critical Care, Pulmonary & Sleep Associates, PLLP/CCT Research, Lakewood, Colorado
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Health Awareness, LLC, Jupiter, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - DelRicht Research, Atlanta, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Optimal Research, LLC, Peoria, Illinois
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - Velocity Clinical Research - Sioux City, Sioux City, Iowa
  - Johnson County Clin-Trials, Lenexa, Kansas
  - DelRicht Research, Louisville, Kentucky
  - IMA Clinical Research, Monroe, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - Profound Research LLC, Clarkston, Michigan
  - Profound Research LLC, Farmington Hills, Michigan
  - Profound Research LLC, Rochester Hills, Michigan
  - DelRicht Research, Gulfport, Mississippi
  - DelRicht Research, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Velocity Clinical Research - Norfolk, Norfolk, Nebraska
  - Velocity Clinical Research - Omaha, Omaha, Nebraska
  - Velocity Clinical Research - Albuquerque, Albuquerque, New Mexico
  - IMA Clinical Research, New York, New York
  - DelRicht Research, Charlotte, North Carolina
  - Velocity Clinical Research - Cleveland, Beachwood, Ohio
  - Velocity Clinical Research - Springdale, Cincinnati, Ohio
  - DelRicht Research, Tulsa, Oklahoma
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Velocity Clinical Research - Anderson, Anderson, South Carolina
  - DelRicht Research, Charleston, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - DelRicht Research, Hendersonville, Tennessee
  - Zenos Clinical Research, Dallas, Texas
  - Lonestar Clinical Research, LLC, Dallas, Texas
  - DelRicht Research, Prosper, Texas
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas
  - Stephenville Medical & Surgical Clinic, Stephenville, Texas
  - Alliance for Multispecialty Research, LLC, Layton, Utah
  - Velocity Clinical Research - Salt Lake City, West Jordan, Utah
  - Clinical Research Partners, LLC, Richmond, Virginia
- hVIVO, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No